CLINICAL TRIAL: NCT05831098
Title: Evaluation of the Sensitivity, Specificity, and Utility of the Reveal® TP (Syphilis) Antibody POCT to Diagnose Infectious Syphilis in Participants Attending the BCCDC's STI Clinic in Vancouver, BC
Brief Title: Evaluation of the Sensitivity, Specificity, and Utility of the Reveal® TP (Syphilis) Antibody POCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedMira Laboratories Inc. (Industry)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MM062TP2022
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Syphilis Infection; Syphilis; Early Syphilis, Symptomatic
Keywords: Rapid Vertical Flow (RVF); Reveal TP; Syphilis; POCT; MedMira
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Masking Description: The result of the Reveal TP (Syphilis) Antibody Test will not be revealed to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Diagnostic: Reveal TP (Syphilis) Antibody Test (Experimental): Participants are tested with investigational devices and conventional syphilis serology tests.
  Interventions: Device: Reveal TP (Syphilis) Antibody Test

INTERVENTIONS:
Device: Reveal TP (Syphilis) Antibody Test — All subjects tested with both investigational devices and conventional syphilis serology tests.
  Other Names: Reveal TP

SUMMARY:
This study is to test the Reveal® TP (Syphilis) antibody POCT (MedMira, Inc., Halifax, Nova Scotia) for its performance in an urban STI clinic in Vancouver, British Columbia and compare its performance in parallel with the usual testing method (the gold standard).

DETAILED DESCRIPTION:
This study is to test the Reveal® TP (Syphilis) antibody POCT (MedMira, Inc., Halifax, Nova Scotia) for its performance in an urban STI clinic in Vancouver, British Columbia and compare its performance in parallel with the usual testing method (the gold standard).

The healthcare professional will advise patients about the study, and with their permission refer them to research staff for recruitment. Should patients choose to participate in the study they will be asked to provide consent to have a few drops of blood sample obtained through a finger prick to be used in the POCT. POCT results will not be provided to participants and this will be explained in both the recruitment script and informed consent form. A sample of 5 to 10 ml venous whole blood will also be obtained for the conventional syphilis serology testing which is part of the routine for care of the four categories of patients (regardless of this research). This research will take approximately 15 to 30 minutes and will be on top of the regular care that patients will receive in the clinic. Upon completing the tests, participants will be asked to complete a brief feedback survey to assess patients' acceptability of syphilis POCT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 19 years of age and above attending the BCCDC STI Clinic in Vancouver, British Columbia for routine sexual health care and requiring syphilis testing as part of this care are eligible for this study.

  * Additionally, for each participant category:

    * Group 1: No known (i.e. self-reported or laboratory documented history of syphilis) prior history of syphilis.
    * Group 2: No additional inclusion criteria
    * Group 3: Participants were named as a contact by a confirmed syphilis case within the last year, and have not yet received treatment
    * Group 4: No additional inclusion criteria
  * Those who had other STIs in the past or being suspected of having other STIs are not excluded as long as testing for syphilis is part of the care provided to them. Once it has been determined that the exclusion criteria does not apply to a patient, the recruitment of the four categories of participants will be offered without other pre-selection criteria unless there may be other unforeseeable circumstances arising, such as shortage of clinic staff or large number of patients showing up.

Exclusion Criteria:

* • Minors, and those who, at the discretion of the health care provider/research co-ordinator, appear intoxicated and/or with extreme distress, or confused, will be excluded from this research because they would not be able to provide informed consent to participate.

  * Additionally, for each participant category:

    * Group 1: Current symptoms that could be consistent with early syphilis.
    * Group 2: No additional exclusion criteria
    * Group 3: Current symptoms that could be consistent with early syphilis.
    * Group 4: Current symptoms that could be consistent with early syphilis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of Reveal TP (Syphilis) Antibody Test | 1 patient visit of approximately 30 minutes
  For each enrolled subject, Reveal TP (Syphilis) Antibody Test will be used to test fingerstick whole blood from the patient. A venipuncture whole blood sample will also be drawn from the patient and will be tested using conventional serological testing methods to determine patient status.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Grennan, Dr, Principal Investigator — British Columbia Center for Disease Control (BCCDC); Raymond Tsang, Dr, Principal Investigator — National Microbiology Laboratory Branch, Public Health Agency of Canada
Locations (1):
- BCCDC STI Clinic, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No